CLINICAL TRIAL: NCT04746404
Title: Application of a Positive Psychology Program for the Development of Emotional Skills in Prison : Feasibility Study
Brief Title: Application of a Positive Psychology Program for the Development of Emotional Skills in Prison
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0017
Record Dates: First submitted 2021-01-29; First posted 2021-02-09 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Control group : Major borderline patients followed up at the Health Unit of the Villeneuve-lès-Maguelone Remand Prison
- Test group: Test group : Major borderline patients followed up at the Health Unit of the Villeneuve-lès-Maguelone Remand Prison
  Interventions: Behavioral: Emotional Skills Development Program

INTERVENTIONS:
Behavioral: Emotional Skills Development Program — Emotional Skills Development Program (positive psychology)
  Groups: Test group

SUMMARY:
Studies show that emotional competence plays a significant role in psychological and physical health, and that programs aimed at their development are effective. Can a positive psychology program aimed at the development of emotional competence be implemented as part of care in lieu of deprivation of liberty? The investigators hypothesize the interest and possibility of implementing an emotional skills development program in the specific context of custodial care.

The main expected outcome of this study is the identification of necessary adaptations of the emotional skills development program of Kotsou, I. et al (2011) for its implementation in remand homes.

DETAILED DESCRIPTION:
The expected secondary outcome is the identification of the interest of emotional skills development program (in prison) regarding :

* Therapeutic support for patients meeting the criteria for borderline personality disorder
* Participant satisfaction
* The development of emotional skills

ELIGIBILITY:
Inclusion criteria:

* Meet the criteria for borderline personality disorder (DSM-V),
* Interest in the issue of emotional skills development,
* Comprehension and use of the French language adapted to the study,
* Disposition to group practice,
* Attentive disposition allowing to participate in a therapeutic activity for 3 hours.
* Psychological/psychiatrical follow-up at the Health Unit of the Villeneuve-lès-Maguelone prison

Exclusion criteria:

* Minor patients
* Releasable before July 2021,
* Decompensated psychiatric disorders,
* Patient in withdrawal syndrome.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patients followed up at the Health Unit of the Villeneuve-lès-Maguelone Remand Prison
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
rate of vompliance with the number of sessions | 1 day
  Achievement of the program's implementation and participation objectives : compliance with the number of sessions
Rate of respect of the frequency of sessions | 1 day
  Achievement of the program's implementation and participation objectives : respect of the frequency of sessions: weekly
rate of respect of the duration of each session | 1 day
  Achievement of the program's implementation and participation objectives : respect of the duration of each session
rate of respect of the minimum number of participants | 1 day
  Achievement of the program's implementation and participation objectives : respect of the minimum number of participants

SECONDARY OUTCOMES:
Respect of the duration of the theoretical/practical reminders | 1 day
  Achievement of the program's implementation and participation objectives : Respect of the duration of the theoretical/practical reminders
respect of the frequency of theoretical/practical remote reminders | 1 day
  Achievement of the program's implementation and participation objectives : respect of the frequency of theoretical/practical remote reminders

CONTACTS AND LOCATIONS:
Overall Officials: Magali RUBIO, Psychologist, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC